CLINICAL TRIAL: NCT04791891
Title: The Quebec Low Back Pain Study (QLBPS): A Platform for the Continuous Enrolment and Longitudinal Epidemiological Evaluation of Individuals With LBP.
Brief Title: Quebec Low Back Pain Study: Core Dataset
Acronym: QLBPS
Status: Recruiting | Type: Observational
Sponsor: Laval University (Other)
Collaborators: Quebec Pain Research Network (Other); Réseau provincial de recherche en adaptation réadaptation (Unknown)
Responsible Party: Sponsor
Other Study IDs: A06-M22-18A
Record Dates: First submitted 2021-03-04; First posted 2021-03-10 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2021-03

CONDITIONS: Low Back Pain
Keywords: Acute; Chronic; Persistence; Inception cohort; Two-stage sampling
MeSH Terms: conditions — Low Back Pain; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Low Back Pain (LBP): Adult women and men with self-reported LBP.
  Inclusion Criteria for potential LBP participants
  * At least 18 years old;
  * Internet access;
  * Fluent in English or French;
  * Self-reported LBP.
  Exclusion Criteria: No exclusion criteria will be adopted in this study.
  * No exclusion criteria will be adopted in this study

SUMMARY:
Persistent back pain is the leading cause of years lived with disability worldwide. Current therapeutic interventions are often either not effective or are associated with undesired consequences. These concerns are further amplified by the current opioid epidemic, resulting in an enormous public health crisis. Experts from diverse disciplines including molecular/cellular biology, neuroscience, psychology and public health formed the Quebec Back Pain Consortium to address this challenge. The overall goal of this project is to facilitate research on factors that contribute to the persistence and recovery from back pain. To accomplish this goal, we will recruit individuals suffering from acute and chronic low back pain across the province of Quebec and follow their pain trajectories over two years using an online platform. During that period, satellite projects will investigate specific risk factors including genetics, diet and physical activity, and advanced statistical methods will be used to integrate and interpret the data. A better understanding of factors influencing back pain will eventually allow for improved early intervention, interruption and prevention.

DETAILED DESCRIPTION:
Introduction The neurobiological mechanisms underlying recovery from or persistence of low back pain (LBP) remain misunderstood, limiting progress towards effective management.

We have developed an innovative two-tier design to study the transition from acute to chronic LBP. The objective of the first tier is to create a provincial web-based infrastructure to recruit and monitor the trajectory of individuals with acute LBP. The objective of the second tier is to fuel hypothesis-driven satellite data collection centers with specialized expertise to study the role of biomechanical, epigenetic, genetic, neuroanatomical, ontological, physiological, psychological, and socioeconomic factors in LBP chronicity.

Methods Adults with acute and chronic LBP will be recruited through networks, media and health care settings. A web-based interface will be used to collect self-reported variables at baseline and at 3, 6, 12 and 24 months. Acute LBP will be defined according to the Dionne 2008 consensus, while chronic LBP will be defined according to Deyo 2014. Measurements will include the Canadian minimum dataset for chronic low back pain research, DN4 for neuropathic pain, comorbidities, EQ-5D-5L for quality of life, and linkage with provincial medico-administrative databases. The primary outcome will be the transition to chronic LBP for the adults with acute LBP at baseline. Secondary outcomes (for both adults with acute and chronic LBP at baseline) include healthcare resource utilization, disability, sick leave, mood, and quality of life. This study brings together diverse research expertise to investigate the transition from acute to chronic LBP, characterize the progression to recovery or chronicity, and identify patterns associated with that progression.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old;
* Internet access;
* Fluent in English or French;
* Self-reported LBP. Presence of LBP will be based on the recommendations of the Standardized Delphi Definitions of Low Back Pain Prevalence. According to these recommendations, LBP is present if both the following questions are answered "yes": (1) In the past 4 weeks, have you had pain in your low back? (2) If yes, was this pain bad enough to limit your usual activities or change your daily routine for more than one day?

Exclusion Criteria:

- No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female, Male, Other
Study Population: The QLBPS will enroll adult women and men with self-reported LBP. The proposed cohort study will be population-based including individuals from urban, remote and rural areas and will not be restricted to patients consulting healthcare professionals substantially improving the generalisability of the results. Potential participants have to be at least 18 years, have internet or phone access, be fluent in either French or English, and have self-reported acute low back pain.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Chronicity: Number of participants who transition from acute to chronic LBP | 6 months
  Chronic LBP will be defined based on the NIH task force recommendations which define chronic LBP as an ongoing problem for at least 3 months and that has resulted in a problem on at least half of the days in the past 6 months.

SECONDARY OUTCOMES:
Work status: number of participants on sick leave | 6 months
  As measured by the self-reported core dataset questionnaire, which includes 2 questions on LBP-related workplace absenteeism and benefits.
Functional limitations: level of function | 6 months
  As measured by the self reported core dataset questionnaire, which includes 4 questions on functional limitations from the Patient-Reported Outcomes Measurement Information System (PROMIS). The level of function is measured on a scale of ''without any difficulty/with little difficulty/ with some difficulty/with much difficulty/'unable to do''. A higher score indicates better outcome.
Health-related quality of life: European Quality of Life Five Dimension Five Level Scale (EQ-5D-5L) score | 6 months
  The EQ-5D-5L score measures five dimensions of health (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) scored on five levels (no, slight, moderate, severe, extreme problems/unable to). A higher score indicates worse outcome (min = 5, max = 25).
Global impression of change of participants' conditions | 6 months
  As measured by the self-reported core dataset questionnaire. Participants rate the extent to which they feel their condition has changed in terms of pain symptoms, functioning and quality of life, in the past 3 months, using a 7-point Likert scale Patient Global Impression of Change (PGIC) (no change / almost the same / a little better / somewhat better / moderately better / better / a great deal better). A higher score indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Sebastien Roy, PhD, PT, Principal Investigator — Laval University
Locations (1):
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/91/NCT04791891/Prot_000.pdf